CLINICAL TRIAL: NCT06035822
Title: Assessment of Nursing Students' Performance During Guided Debriefing With the Lasater Clinical Judgement Rubric: a Randomized Clinical Trial
Brief Title: Assessment of Nursing Students' Performance During Guided Debriefing With the Lasater Clinical Judgement Rubric
Acronym: SIM_LCJR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vic - Central University of Catalonia (Other)
Responsible Party: Principal Investigator, Montserrat Faro, Principal investigator Dr. Montserrat Faro-Basco, University of Vic - Central University of Catalonia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: SIM_DEB_LCJR
Record Dates: First submitted 2023-09-06; First posted 2023-09-13 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-11

CONDITIONS: Educational Activities

STUDY DESIGN:
Intervention Model Description: The assignment of the 30 groups to the intervention or control group was randomized. Fifteen were assigned to the intervention group (IG) and were given the High-Fidelity Simulation (HFS) intervention with a debriefing script, and 15 were assigned to the control group (CG) and were given the HFS intervention without a debriefing script.
Who Masked: Participant, Outcomes Assessor
Masking Description: The students did not know whether they were a control group or an intervention group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Debriefing with TeamGAINS (Experimental): The Intervention Group debriefings (n=15) were conducted by the research teacher, who is trained in clinical simulation methodology, is a clinical simulation instructor, and is trained in the use of the TeamGAINS tool (Kolbe et al., 2013).
  The intervention consisted of using the TeamGAINS tool as a debreifing script, during the debriefing, in accordance with the objectives of the clinical simulation scenario (CSC).
  Interventions: Other: Debriefing with TeamGAINS
- Debriefing free (No Intervention): The Control Group debriefings (n=15) were conducted by a teacher trained in clinical simulation methodology, with no experience in the use of any debriefing guide.
  The intervention consisted of the debriefer applying his or her simulation experience and training to perform the debriefings freely, in accordance with the objectives of the clinical simulation scenario (CSC).

INTERVENTIONS:
Other: Debriefing with TeamGAINS — The IG debriefings were conducted by the research teacher, who is trained in clinical simulation methodology, is a clinical simulation instructor, and is trained in the use of the TeamGAINS tool, using this tool as a debriefing script, in accordance with the objectives Clinical Simulation Scenario
  Arms: Debriefing with TeamGAINS

SUMMARY:
I invite you to participate in the study entitled Use of debriefing as a training tool in simulation, of which Montserrat Faro-Basco is not the main researcher. The study is linked to the doctoral thesis Debriefing in clinical simulation, essential for the development of reflective professionals, which the same researcher is carrying out as part of the UVic-UCC Doctoral Program in Educational Innovation and Intervention.

The aim of this study is:

- Analysis of the effectiveness of the structured debriefing session with the TeamGAINS tool

The procedure to follow will consist of the recording of the debriefing for the subsequent analysis of the behaviors and attitudes of the participants in the session (teacher and students), through its viewing.

Participation in this activity is voluntary and does not involve any harm or danger to your physical or mental health. You can refuse to participate at any time in the study without having to give reasons for this, or receiving any type of penalty.

The data obtained will be confidential, anonymity will be kept, these data will be organized with a number assigned to each participant, there will be no record of the identity of the participants. The data will be in charge of the research team of this study for the subsequent development of reports and publications of the study results in scientific journals.

The collected information will not be used for any purpose other than those indicated.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criterion applied was all students enrolled in the Practicum VI subject in the 2017-2018 academic year.

Exclusion Criteria:

* The exclusion criterion was students who did not wish to participate in the study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Number of participants who have improved their performance from structured debriefing and good clinical reasoning. | The evaluation instrument is applied during the debriefing analysis carried out at the end of the intervention, lasting one hour.
  The debriefing sessions were recorded with two fixed video cameras, which were activated at the beginning of the debriefing. The purpose of the recordings was that the two facilitators and the two external evaluators could later view them in order to be able to analyze and evaluate the participants' interventions during the debriefing, applying the LCJR instrument, which allowed the assessment of the student's performance and clinical reasoning.

CONTACTS AND LOCATIONS:
Locations (1):
- c. Sagrada Familia, 7, Vic, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided